CLINICAL TRIAL: NCT05418660
Title: Observational Retro-prospective Study on Programmed Cell Death 1/ Programmed Cell Death Ligand1 (PD1/PDL1) Inhibitors Treatment Duration in Patients With Non Small Cell Lung Carcinoma
Brief Title: Observational Retro-prospective Study on PD1/PDL1 Inhibitors Treatment Duration in Patients With NSCLC
Acronym: I-STOP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milano Bicocca (Other)
Collaborators: Azienda Ospedaliera San Gerardo di Monza (Other)
Responsible Party: Sponsor
Other Study IDs: I-STOP
Record Dates: First submitted 2022-05-27; First posted 2022-06-14 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Immunotherapy; nivolumab; atezolizumab; pembrolizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immunotherapy; Nivolumab; pembrolizumab; atezolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: The cohort includes patients who discontinue the treatment at 24 months and continue the follow-up at least for 3 months
  Interventions: Drug: Immunotherapy
- Cohort 2: The cohort includes patients who continue the treatment beyond 24 months until unacceptable toxicity or progression.
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Drug: Immunotherapy — At least 24 months with Pembrolizumab, Nivolumab or Atezolizumab in any treatment line
  Other Names: Nivolumab; Pembrolizumab; Atezolizumab

SUMMARY:
Retrospective/ prospective, multicentre, international observational study on long-responders with non-small cell lung carcinoma patients treated with anti Programmed cell Death 1/ Programmed cell Death Ligand 1 (anti-PD1/PD-L1) in any line of treatment for at least 24 months with response partial/complete response or disease stability. Patients will be divided into two cohorts based on whether they stopped treatment at 24 months (not for toxicity) or continued by clinical choice and stratified according to treatment line and baseline PD-L1 expression.

DETAILED DESCRIPTION:
Programmed cell Death protein / Ligand 1 (PD-1 / PD-L1) inhibitors Atezolizumab, Nivolumab and Pembrolizumab have demonstrated a great efficacy and a good safety profile in patients with Non-Small Cell Lung Cancer (NSCLC), both in first-line (PD-L1 expression > 50%) and in subsequent lines regardless of PD-L1 status. Recently, the combination of Pembrolizumab with platinum salts and pemetrexed has become the gold standard for the first-line treatment in patients with PD-L1 expression <50%. Data on the optimal duration of immunotherapy are scarce, especially considering that the onset of immune-related adverse events (irAE) has also been reported after several months of treatment and the long-term effects of the persistent immune system stimulation are unknown. Furthermore, predictive factors are not available to identify those patients who will respond to treatment and could benefit from a shorter duration of therapy -this information is pivotal to minimize the risk of side effects and improve the quality of life. Basal characteristics, such as PD-L1 expression, percentage of Cluster of Differentiation 8 (CD-8) + T-lymphocyte in tumor-infiltrating lymphocytes (TILs), mutational status, neutrophil to lymphocyte ratio (NLR), and platelets to lymphocytes ratio (PLR) have been reported as possible biomarkers, but further data are needed to confirm their predictive value. The purpose of the study is to identify the differences in terms of effectiveness and safety of immunotherapy in long-responder patients in the two cohorts. Secondary objectives are to evaluate the outcome after anti-PD1/PD-L1 rechallenge or other treatment for patients who progress after immunotherapy discontinuation and to identify baseline characteristics that may be predictive of response (molecular characteristics, biohumoral parameters, body mass index).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically / cytologically confirmed diagnosis of NSCLC, with or without brain metastases
3. Illness measurable according to Response Evaluation Criteria in Solid Tumours (iRECIST) criteria
4. At least 24 months of treatment with Pembrolizumab, Nivolumab or Atezolizumab
5. Complete response (CR)/ partial response (RP)/ stable disease at the end of 24-month treatment. The maintenance of the response may also have been obtained after loco-regional treatment, e.g. surgery or radiotherapy, in the case of oligoprogression for a maximum of 3 locoregional treatments (e.g. radiotherapy, surgery) throughout the period of treatment and suspension. Even progression at the brain level, treated with radiation therapy or surgery, can be considered, provided that it is followed by a disease control for at least 3 months.
6. At least 3 months of follow-up or death within three months after stopping the 24-month treatment.
7. Informed consent freely granted and acquired before the start of the study, for alive and contactable patients.

Exclusion Criteria:

1. Initial chemo-immunotherapy treatment or association with other immunotherapy or other drugs in the context of clinical trials.
2. Permanent discontinuation of treatment with anti PD-1 / PD-L1 for adverse events.
3. More than 3 loco-regional treatments for maintaining the radiological response
4. Suspension of immunotherapy for a period longer than 40 days during the 24-month treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of NSCLC patients treated for at least 24 months with Pembrolizumab, Nivolumab or Atezolizumab in any treatment line. The patients should obtain and maintain a partial (RP) or complete response (RC) or stable disease (SD) at the end of the 24-month therapy.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free survival | Through study completion, an average of 18 months
  Progression free survival (PFS) in the two cohorts; at least 24 months with Pembrolizumab, Nivolumab or Atezolizumab in any treatment line
Overall survival | Through study completion, an average of 18 months
  Overall survival (OS) in the two cohorts; OS will be calculated from the first day of treatment until the date of death from any cause.
Percentage of patients with disease progression after 24 months of treatment | Through study completion, an average of 18 months
  Proportion of patients who show disease progression according to Response Evaluation Criteria in Solid Tumours (RECIST) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Diego Cortinovis, MD, Principal Investigator — Fondazione IRCCS San Gerardo dei Tintori, Monza
Locations (10):
- Italy (10):
  - AOU Ospedali Riuniti, Ancona
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale Policlinico San Martino, Genova
  - Azienda Ospedaliero Universitaria, Modena
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Istituto Nazionale dei Tumori, Napoli
  - Azienda Ospedaliero Universitaria San Luigi, Orbassano
  - Azienda Ospedaliero Universitaria, Parma
  - Azienda Ospedaliera Marche Nord, Pesaro
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine

IPD SHARING:
Plan to Share IPD: No
Data will be available upon request